CLINICAL TRIAL: NCT01058044
Title: A Pilot Study of Adherence to Oral Anticancer Treatment Using Electronic Monitoring System
Brief Title: Adherence to Oral Anticancer Treatment Using Electronic Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AU792; RCB 2009-A00244-53 (Other: France: Afssaps - French Health Products Safety Agency)
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Cancer
Keywords: Cancer, Sunitinib, capecitabine, anastrozole, letrozole; adherence, anticancer treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adherence assessment group (Experimental): evaluation of adherence using MEMS
  Interventions: Other: Evaluation of adherence to 3 oral anticancer treatment using a " Medication Event Monitoring System "

INTERVENTIONS:
Other: Evaluation of adherence to 3 oral anticancer treatment using a " Medication Event Monitoring System " — Evaluation of adherence using a " Medication Event Monitoring System " (MEMS®) for oral anticancer treatment delivered by dispensary pharmacy

SUMMARY:
The purpose of this study is to describe adherence to 3 oral anticancer treatment: i) a chemotherapeutic regimen with capecitabine (alone or in association with lapatinib), ii) or sunitinib an tyrosine kinase inhibitor, iii) or an non-steroidal aromatase inhibitor. Moreover, this study is aimed at evaluating the feasibility to use a " Medication Event Monitoring System " (MEMS®) in order to assess adherence of an oral anticancer treatment delivered by dispensary pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* histologically proven malignant tumor
* documented decision of treatment with i) a chemotherapeutic regimen with capecitabine (alone or in association with lapatinib), ii) or sunitinib an tyrosine kinase inhibitor, iii) or an non-steroidal aromatase inhibitor
* ambulatory treated subject
* Subject who accept to use MEMS monitors to automatically compile their drug dosing histories
* Written informed consent

Exclusion Criteria:

* any severe concomitant wich makes it undesirable for the patient to participate in the study or which would jeopardize adherence with trial protocol
* patient who does not agreed to participate the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
evaluation of adherence to 3 oral anticancer treatment: i) a chemotherapeutic regimen with capecitabine (alone or in association with lapatinib), ii) or sunitinib an tyrosine kinase inhibitor, iii) or an non-steroidal aromatase inhibitor. | everey visit during 6 months

SECONDARY OUTCOMES:
evaluation of liberal nurse satisfaction | inclusion
resort to healthcare system (oncologist, doctor, nurse, hospital pharmacy, dispensary pharmacy) | during 6 months
Patient satisfaction | 6 months
drug interaction | during 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France